CLINICAL TRIAL: NCT03541577
Title: Sensor-equipped Ultrathin Pressure Microcatheter Versus Pressure Wire for FFR Measurement: A Multi-center Prospective Control Study
Brief Title: Sensor-equipped Ultrathin Pressure Microcatheter Versus Pressure Wire for FFR Measurement
Acronym: SUPREME
Status: Completed | Type: Observational
Sponsor: Insight Lifetech Co., Ltd. (Industry)
Collaborators: Shanghai Zhongshan Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); Guangdong Provincial People's Hospital (Other); Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CTP17-001
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Coronary Disease; Myocardial Ischemia
MeSH Terms: conditions — Coronary Artery Disease; Coronary Disease; Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants: Subjects who meet the inclusion criteria and do not meet the exclusion criteria and undergo FFR measurement with the TruePhysioTM Microcatheter and the Pressure Wire
  Interventions: Device: TruePhysioTM Microcatheter; Device: Pressure Wire

INTERVENTIONS:
Device: TruePhysioTM Microcatheter — Provide hemodynamic information for the diagnosis and treatment of coronary and peripheral artery disease. The system is intended for use in catheterization and related cardiovascular specialty laboratories to compute and display fractional flow reserve (FFR).
  Other Names: FFR Microcatheter
Device: Pressure Wire — Provide hemodynamic information for the diagnosis and treatment of coronary and peripheral artery disease. The system is intended for use in catheterization and related cardiovascular specialty laboratories to compute and display fractional flow reserve (FFR).
  Other Names: PressureWire

SUMMARY:
TruePhysioTM Sensor-equipped Ultrathin Pressure Microcatheter (referred to as TruePhysioTM Microcatheter below) is a novel device for evaluating the functional significance of coronary stenosis. This study will compare the differences, if any, between the coronary fractional flow reserve (FFR) measured by the TruePhysioTM Microcatheter and the Pressure Wire.

DETAILED DESCRIPTION:
Many studies have reported that FFR-guided coronary revascularization leads to improved long-term clinical outcomes and reduced costs compared with angiography-guided coronary revascularization alone. Current guidelines emphasize the measurement of FFR as the standard of reference when determining the functional significance of coronary artery stenosis in stable patients when evidence of ischemia is not available (class IA indication). But FFR is still underutilized in clinical practice. One of the reasons may be the difficulty in manipulating the Pressure Wire.

TruePhysioTM Microcatheter is a novel device for evaluating the functional significance of coronary stenosis, which may simplify FFR measurements by allowing the use of standard guidewires best suited to negotiating the patients' anatomy. This study is a prospective, open label, multi-center study with the purpose of comparing the differences, if any, between FFR measured by the TruePhysioTM Microcatheter and Pressure Wire. The secondary purpose is to analyze the correlation between FFR measured by the TruePhysioTM Microcatheter and Pressure Wire. A total of 239 patients will be recruited at 4 centers in China.

ELIGIBILITY:
General Inclusion Criteria:

* Age: 18-75 years old
* Subjects with coronary artery disease
* Able to understand and provide signed consent

Angiographic Inclusion Criteria:

* Subject has an intermediate stenosis in a native coronary vessel
* The target stenosis has a reference diameter ≥2.50 mm by visual assessment.

Exclusion Criteria:

General Exclusion Criteria:

* Acute ST-elevation or non-ST-elevation myocardial infarction
* Severe heart failure (NYHA≥IV)
* Left ventricular ejection fraction <30%
* Allergy to adenosine triphosphate (ATP)
* Contraindications for percutaneous coronary intervention (PCI)

Angiographic Exclusion Criteria:

* Target vessel has angiographically visible or suspected thrombus
* Angiographic evidence of a dissection
* Excessive tortuosity or calcification stenosis, left main stenosis, serial stenosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease for whom FFR measurement is thought to be clinically indicated.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
FFR Measurements | Duration of FFR measurement
  Comparisons between the FFR measured by the TruePhysioTM Microcatheter and the Pressure Wire (PW), including bias, as assessed by Bland-Altman analysis.

SECONDARY OUTCOMES:
Pearson analysis | Duration of FFR measurement
  Pearson analysis of paired FFR measurements by TruePhysioTM Microcatheter and PW.
Slope of Passing-Bablok fit | Duration of FFR measurement
  Slope of Passing-Bablok fit between paired FFR measurements by TruePhysioTM Microcatheter and PW.
Intercept of Passing-Bablok fit | Duration of FFR measurement
  Intercept of Passing-Bablok fit between paired FFR measurements by TruePhysioTM Microcatheter and PW.
Diagnostic FFR concurrence of functionally significant stenosis | Duration of FFR measurement
  Concurrence of TruePhysioTM Microcatheter FFR diagnostic accuracy of functionally significant stenosis, using PW FFR ≤0.80 as the reference.
Sensitivity, Specificity of TruePhysioTM Microcatheter in determining functionally significant stenosis | Duration of FFR measurement
  Sensitivity, Specificity of TruePhysioTM Microcatheter in determining functionally significant stenosis at the vessel level with PW FFR as the reference standard (PW FFR ≤0.80 as positive case).
Device success rate | Duration of FFR measurement
  Device success rate, defined as a valid FFR reading for each system, and comparison between the two systems.
Mean drift | Duration of FFR measurement
  Mean drift, defined as the absolute difference between Pd/Pa at the equalization position after pullback and 1.00, for each system, and comparison between the two systems.
Rate of clinically significant drift | Duration of FFR measurement
  Rate of clinically significant drift (drift >0.03), for each system, and comparison between the two systems.
Rate of device-related adverse effects | Duration of FFR Procedure
  Rate of device-related adverse effects, for each system individually, and comparison between the two systems.
PW FFR measurements with TruePhysioTM Microcatheter across and not across lesion | Duration of FFR Procedure
  Comparisons between PW FFR measurements with TruePhysioTM Microcatheter across lesion and with TruePhysioTM Microcatheter not across lesion, including bias, as assessed by Bland-Altman analysis.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Guangdong General Hospital, Guangzhou
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou
  - Shanghai Zhongshan Hospital, Shanghai
  - Shenzhen People's Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li C, Yang J, Dong S, Dong L, Chen J, Shen L, Zhang F, Li C, Liu H, Hu X, Hau WK, Qian J, Jeremias A, Wang J, Ge J; SUPREME Study Investigators. Multicenter clinical evaluation of a piezoresistive-MEMS-sensor rapid-exchange pressure microcatheter system for fractional flow reserve measurement. Catheter Cardiovasc Interv. 2021 Aug 1;98(2):E243-E253. doi: 10.1002/ccd.29678. Epub 2021 May 5. PMID 33951285